CLINICAL TRIAL: NCT00669656
Title: A Phase II Trial of a Combination Herbal Therapy for Men With Biochemical Recurrence of Prostate Cancer After Initial Local Therapy
Brief Title: Herbal Therapy for Treatment of Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-07-3
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cholecalciferol; alpha-Tocopherol; Vitamin E; Selenium; Tea; gallocatechol; saw palmetto extract; Lycopene; daidzein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prostate Health Cocktail (Experimental)
  Interventions: Drug: Prostate Health Cocktail

INTERVENTIONS:
Drug: Prostate Health Cocktail — 3 capsules daily PO up 12 months
  Other Names: Cholecalciferol; Vitamin D3; d-alpha tocopherol; vitamin E; L-selenomethionine; selenium; green tea extract; EGC; Epigallocatechin; saw palmetto; lycopene; Isoflavanoids; Daidzein; Genisetein

SUMMARY:
This study is about Prostate Health Cocktail, a combination supplement that contains vitamin D3, vitamin E, selenium, green tea extract, saw palmetto, lycopene, and soy derivatives. This product is currently available on the market, as herb and vitamin supplements are not regulated by the FDA. Each ingredient has been studied in prostate cancer cells and/or in patients with prostate cancer. At the doses included in this supplement, no serious side effects have been reported.

The purpose of this study is to find out whether Prostate Health Cocktail can lower your PSA. Additionally, we will be looking to see whether taking this treatment causes any unexpected side effects, and whether certain blood tests can inform us about your disease status in addition to your PSA

DETAILED DESCRIPTION:
Objectives of this study are:

* To assess the PSA response in prostate cancer patients who have a PSA-only disease recurrence after curative local therapy, during treatment with a combination herbal supplement.
* To qualitatively and quantitatively describe the toxicity profile of this herbal supplement.
* To assess changes in PSA doubling time for subjects treated with this supplement.
* To measure tissue GRP78, serum neuroendocrine markers, and circulating tumor cells, for correlation with treatment response and prostate cancer outcomes

ELIGIBILITY:
Inclusion Criteria::

* Age greater than or equal to 18
* Histologically documented adenocarcinoma of the prostate
* Initial treatment with radical prostatectomy or external beam radiation

  * Neoadjuvant/Adjuvant Androgen Deprivation therapy allowable, provided it was for a maximum of 24 months, with the last dose of medication at least 12 months previously
  * Neoadjuvant or adjuvant chemotherapy allowable, provided it was for a maximum of 6 months, with the last dose of medication at least 12 months previously
  * Adjuvant radiation after radical prostatectomy is allowed, provided at least 6 months have elapsed between completion of radiation and enrollment in study
* PSA recurrence, with a rising PSA, as defined by:

  * Post Radiation Therapy:

    * Absolute PSA >2.0 ng/mL
    * PSA nadir <4 ng/mL after radiation
    * Absolute rise of at least 0.5 ng/mL total
    * At least 2 increases in PSA, separated by at least 2 weeks; these can be separated by a PSA value which declines provided the second rising value is higher than the first rising value.
  * Post Prostatectomy:

    * Absolute PSA >1.0 ng/mL
    * Absolute rise of at least 1 ng/mL total from nadir
    * At least 2 increases in PSA separated by at least 2 weeks; these can be separated by a PSA value which declines provided the second rising value is higher than the first value
* PSA Doubling Time (PSA DT) more than 3 months and less than 36 months

  * PSA DT to be calculated using the web-based calculator at http://kevin.phys.unm.edu/psa/ with the following constraints:

    * At least 3 values, but no more than 6
    * All values must be >0.2
    * Values must be separated by at least 2 months
* No radiographically evident bony or soft tissue metastases
* Documented discussion between subject and physician about the option to pursue hormone therapy and/or salvage local therapy rather than enroll in this study
* Patients who received treatment with androgen deprivation for biochemical recurrence are eligible provided:

  * They did not document castration resistance (defined as 2 rising PSA values while testosteron < 50
  * They have been off androgen deprivation for at least 3 months and have recovered their testosterone (>150)
  * They have decided,in conjunction with their treating physician that they do not want to resume androgen deprivation
* ECOG Performance Status 0-2
* Life expectancy > 12 months
* Adequate hepatic function (AST, ALT, bilirubin <1.5 x ULN)
* Adequate renal function (eGFR by Cockcroft-Gault or comparable calculation >50 ml/min)
* Willing to discontinue all nutritional supplements and 5-alpha reductase inhibitors (finasteride, dutasteride) for the duration of study treatment, unless the medication is being used to control symptoms of BPH and the patient has been taking the medication for more than 6 weeks
* Willing to discontinue all weight control medications for the duration of study treatment
* Signed informed consent

Exclusion Criteria:

* Atypical prostate carcinoma histology (ex: small cell, adenoid cystic)
* Evidence of bony or soft tissue metastatic disease on CT/MRI or bone scan or PET/CT
* Other invasive malignancy within prior 3 years, except for fully treated basal cell or squamous cell carcinoma of the skin.
* Full-dose anticoagulation therapy (warfarin or low molecular weight heparin) or antiplatelet therapy (clopidogrel or ticlopidine), with the exception of low-dose aspirin therapy (81 mg).
* Significant cardiac disease, included but not limited to angina, myocardial infarction, cardiomyopathy, congestive heart failure, and coronary artery disease which has required bypass surgery, angioplasty or stent placement.
* Significant uncontrolled comorbid condition which, in the opinion of the treating physician would compromise the subject's ability to comply with protocol requirements, or would pose undue risk for experiencing adverse events.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-07-06 (Actual); Primary Completion 2014-07-08 (Actual); Study Completion 2014-10-14 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this trial will be PSA response | PSA measurement every 4 weeks

SECONDARY OUTCOMES:
Toxicity and side effects | Assessed every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Dorff, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States